CLINICAL TRIAL: NCT02475226
Title: Distribution and Mortality Factors of Cases With Traumatic and Non Traumatic Brain Damage Treated in Intensive Care; Retrospective Clinical Trial
Brief Title: Cases With Traumatic and Non Traumatic Brain Damage Treated in the Intensive Care
Status: Completed | Type: Observational
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gulsah Karaoren, MD, Umraniye Education and Research Hospital
Other Study IDs: GK7
Record Dates: First submitted 2015-06-15; First posted 2015-06-18 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Brain Injuries
Keywords: Traumatic Brain Injury; Brain Damage; Mortality; C10.228.140.199
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients with body and head trauma: type of the brain injury in patients with brain damage associated both general body and head trauma
  Interventions: Other: type of the brain injury
- Patients with pure head trauma: type of the brain injury in patients with brain damage associated pure head trauma
  Interventions: Other: type of the brain injury
- Patients with spontaneous hemorrhage: type of the brain injury in Patients with brain damage associated spontaneous hemorrhage
  Interventions: Other: type of the brain injury

INTERVENTIONS:
Other: type of the brain injury — epidural hematoma
Other: type of the brain injury — subdural hematoma
Other: type of the brain injury — subarachnoid hematoma
Other: type of the brain injury — intraparenchymal hematoma
Other: type of the brain injury — scull fracture
Other: type of the brain injury — brain contusion

SUMMARY:
Cases of traumatic and nontraumatic brain damage have high rates of morbidity and mortality. In this study of cases being treated in the ICU for a diagnosis of brain damage, it was aimed to evaluate the relationship between mortality and the distribution of reason for and resulting type of brain damage and to determine other factors affecting mortality.

DETAILED DESCRIPTION:
After local ethics committee approval, a total of 1004 patients treated in the ICU in a 2-year period were retrospectively reviewed. 135 patients, determined with traumatic or nontraumatic brain damage, with a more than 24-hour stay in the ICU, included the study. Reasons for brain damage were determined as brain damage associated with pure head trauma (Group HT), head trauma accompanying general body trauma (Group HT+GBT) and spontaneous haemorrhage (Group SH). The type of brain damage was defined from the radiological diagnosis as subarachnoid haemorrhage, intracranial haemorrhage (ICH), subdural haematoma(SDH), epidural haematoma(EDH), skull fracture, brain contusion or a combination of these (COM).

ELIGIBILITY:
Inclusion Criteria:

* Patients treated in the ICU with the diagnose of traumatic or nontraumatic brain damage, with a more than 24-hour stay.

Exclusion Criteria:

* Patients admitted less than 24 hour.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: a total of 1004 patients treated in the ICU in a 2-year period were retrospectivly reviewed. 135 patients, determined with traumatic or nontraumatic brain damage, with a more than 24-hour stay in the ICU, included the study.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2015-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
number of patients by brain damage types | 2 years
  distribution of the patients with brain damage over the brain damage reasons

SECONDARY OUTCOMES:
Number of factors effecting the mortality | 2 years
  duration time of intubation, duration time in the ICU, APACHE scores, GCS scores.

CONTACTS AND LOCATIONS:
Overall Officials: Nurten Bakan, MD, Study Chair — Umraniye Education and Research Hospital
Locations (1):
- Istanbul Umraniye Education and Research Hospital, Istanbul, Turkey, Turkey (Türkiye)

REFERENCES:
- [Result] Sacco S, Marini C, Toni D, Olivieri L, Carolei A. Incidence and 10-year survival of intracerebral hemorrhage in a population-based registry. Stroke. 2009 Feb;40(2):394-9. doi: 10.1161/STROKEAHA.108.523209. Epub 2008 Nov 26. PMID 19038914
- [Result] Schwarz S, Hafner K, Aschoff A, Schwab S. Incidence and prognostic significance of fever following intracerebral hemorrhage. Neurology. 2000 Jan 25;54(2):354-61. doi: 10.1212/wnl.54.2.354. PMID 10668696